CLINICAL TRIAL: NCT06913088
Title: Ultrasonication-mediated Microbubbles Dressings Increase the Therapeutic Efficacy of Piroxicam Gel for Hand Arthritis: Assessments Using Conventional and Ultrafast Power Doppler Imaging
Brief Title: Ultrasonication-mediated Microbubbles Dressing for Hand Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Kuo-Lung Lai, Doctor, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCVGH-1123802B
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Hand Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBUS group (Experimental): ultrasonication-mediated microbubbles dressing (day 1,3,5) + piroxicam gel (day 2,4,6,7)
  Interventions: Procedure: ultrasonication-mediated microbubbles dressing
- US group (Sham Comparator): ultrasonication using pure gel (day 1,3,5) + piroxicam gel (day 2,4,6,7)
  Interventions: Procedure: ultrasonication using pure gel
- Control group (No Intervention): piroxicam gel alone (day 1-7)

INTERVENTIONS:
Procedure: ultrasonication-mediated microbubbles dressing — The microbubble suspension is diluted with normal saline to a concentration of 2x10^7 bubbles/mL, applied to a gauze cloth, and covered on the joint skin surface. The joint is ultrasonicated for 3 minutes using an ultrasonic implanter (KUM-2000, NEO-TEC, Taipei, Taiwan), and then piroxicam gel is applied. The parameter values for ultrasonication are duty cycle 0.5, Tempo 10, intensity 70%, and time 3 min. This treatment is performed on day 1, 3, and 5.
  Arms: MBUS group
Procedure: ultrasonication using pure gel — The joint is ultrasonicated for 3 minutes using an ultrasonic implanter (KUM-2000, NEO-TEC, Taipei, Taiwan) with pure gel, and then piroxicam gel is applied. The parameter values for ultrasonication are duty cycle 0.5, Tempo 10, intensity 70%, and time 3 min. This treatment is performed on day 1, 3, and 5.
  Arms: US group

SUMMARY:
The goal of this clinical trial is to learn if ultrasonication-mediated microbubbles dressing works to treat hand arthritis in adults. It will also learn about the safety of ultrasonication-mediated microbubbles dressing. The main questions it aims to answer are:

Does ultrasonication-mediated microbubbles dressing increase the therapeutic efficacy of piroxicam gel for hand arthritis?

Researchers will compare "ultrasonication-mediated microbubbles dressing + piroxicam gel " to "ultrasonication + piroxicam gel" and "piroxicam gel alone" to see if ultrasonication-mediated microbubbles dressing works to treat hand arthritis.

Participants will:

Take "ultrasonication-mediated microbubbles dressing (day 1,3,5) + piroxicam gel (day 2,4,6,7) ", "ultrasonication (day 1,3,5) + piroxicam gel (day 2.4.6.7)", and "piroxicam gel alone (day 1-7)" for 1 week.

Visit the clinic on day 1 and day 8 for checkups and tests Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hand arthritis
* Have at least three symptomatic joints over wrist, metacarpophalangeal joints, and interphalangeal joints

Exclusion Criteria:

* Infectious arthritis
* Acute gout

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response | day 8
  A decrease in pain visual analogue scale (VAS) score of ≥2 on day 8 relative to day 1, or an absolute VAS score of ≤1 on day 8.
  [Pain VAS score range: 0-10, higher scores mean a worse outcome]
B-mode response | day 8
  A ≥20% decrease in synovial area on day 8 relative to day 1
Conventional power Doppler (PD) response | day 8
  A ≥20% decrease in synovial PD area on day 8 relative to day 1 on conventional PD image

SECONDARY OUTCOMES:
Ultrafast PD response | day 8
  A ≥20% decrease in synovial PD area on day 8 relative to day 1 on ultrafast PD image

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taichung, Taiwan